CLINICAL TRIAL: NCT01793129
Title: A Randomized Trial of Targeted Temperature Management With Whole Body Hypothermia For Moderate And Severe Hypoxic-Ischemic Encephalopathy In Premature Infants 33-35 Weeks Gestational Age.
Brief Title: Preemie Hypothermia for Neonatal Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0051; U10HD021364 (NIH); U10HD040689 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027904 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD021373 (NIH); U10HD040492 (NIH); U10HD053109 (NIH); U10HD040461 (NIH); U10HD068244 (NIH); U10HD068263 (NIH); U10HD068270 (NIH); U10HD068278 (NIH); U10HD068284 (NIH); U10HD036790 (NIH); UG1HD087226 (NIH)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Results first posted 2024-04-22 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Infant, Newborn; Hypoxia, Brain; Hypoxia-Ischemia, Brain; Encephalopathy, Hypoxic-Ischemic; Hypoxic-Ischemic Encephalopathy; Ischemic-Hypoxic Encephalopathy
Keywords: NICHD Neonatal Research Network; Hypoxic-ischemic encephalopathy (HIE); Hypothermia; Neonatal depression; Perinatal asphyxia
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia-Ischemia, Brain; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Whole-body Hypothermia (Experimental): Induced Whole-body hypothermia (with a target esophageal temperature of 33.5°C) for 72 hours
  Interventions: Device: Hypothermia
- Normothermia (Placebo Comparator): Control group (with esophageal temperature at or near 37.0°C) for 72 hours
  Interventions: Procedure: Normothermic Control

INTERVENTIONS:
Device: Hypothermia — Induced Whole-body hypothermia (with a target esophageal temperature of 33.5°C) for 72 hours
  Arms: Whole-body Hypothermia
Procedure: Normothermic Control — Normothermic Control group (with esophageal temperature at or near 37.0°C) for 96 hours
  Arms: Normothermia

SUMMARY:
This study is a randomized, controlled trial to assess safety and effectiveness of whole body hypothermia for 72 hours in preterm infants 33-35 weeks gestational age (GA) who present at <6 hours postnatal age with moderate to severe neonatal encephalopathy (NE). The study will enroll infants with signs of NE at 18 NICHD Neonatal Research Network sites, and randomly assign them to either receive hypothermia or participate in a non-cooled control group.

DETAILED DESCRIPTION:
Most clinical studies of neonatal encephalopathy (NE) and potential interventions have focused on infants ≥36 weeks GA. Although many interventions have been suggested and assessed for prevention or palliation of NE, the only one currently supported by rigorous clinical evidence to improve outcome in human newborns has been hypothermia implemented at <6 hours of postnatal age and maintained for 72 hrs. Data about diagnosis, frequency, severity, and outcome of NE in infants 33-35 weeks GA are sparse.

This trial will assess safety and effectiveness of whole body hypothermia for 72 hours in preterm infants 33-35 weeks gestational age (GA) who present at <6 hrs postnatal age with moderate to severe neonatal encephalopathy. Infants 33 0/7 to 35 6/7 weeks GA (best obstetrical estimate) and greater than or equal to 1500 grams birth weight (selected to minimize potential difficulties placing esophageal probe) who meet clinical, biochemical and neurologic criteria for moderate to severe NE will be randomized to either whole body hypothermia or participate in a non-cooled control group. The primary outcome will be death or moderate to severe disability at 18-22 months corrected age. The presence or absence of disability will be determined by the standard NRN interdisciplinary follow-up exam.

Secondary Study includes determining an association between MRI detectable injury and neurodevelopment at 18-22 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants 33 0/7 to 35 6/7 weeks GA (best obstetrical estimate)
* Infants weight greater than or equal to 1500 grams at birth
* Postnatal age less than 6 hours
* Infants who meet clinical, biochemical and neurologic criteria for moderate to severe NE:

Biochemical: Cord gas or blood gas within first hour of life with pH ≤7.00 or base deficit (BD) ≥16 mEq/L OR

Acute perinatal event (e.g., abruptio placenta, cord prolapse, uterine rupture, severe FHR abnormality such as variable or late decelerations) AND Requirement for positive pressure ventilation for apnea or poor respiratory effort since birth for at least 10 minutes OR 10 minute Apgar score ≤5

AND

Neurologic:

Seizures OR modified Sarnat score with abnormalities in at least 3 of the 6 categories; at least one must be altered level of consciousness (lethargy or stupor/coma) as determined by a certified examiner (All infants who meet criteria for potential inclusion will undergo standard neurologic exam as for infants ≥36 wks GA being considered for hypothermia, with findings recorded)

Exclusion Criteria:

* Receipt of sedative, analgesic or paralytic agent that may confound the qualifying neurologic exam
* Etiology of NE not likely to be hypoxic-ischemic in origin
* Major congenital anomaly that may confound outcome
* Considered to be moribund and will not be receiving full intensive care
* Equipment and/or appropriate staff not available
* Core temperature < 33.5oC for more than one hour at time of screening
* Unable to randomize by 6 hours of age
* Infant needs ECMO
* All blood gases (cord and postnatal at < 1hr of age) have a pH > 7.15 AND a base deficit < 10mEq/L

Ages: 33 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2015-05; Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele C Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; C. Michael Cotten, MD, Principal Investigator — Duke University; David P Carlton, MD, Principal Investigator — Emory University; Greg Sokol, MD, MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Brenda Poindexter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Wally A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F Bell, MD, Principal Investigator — University of Iowa; Kristi L Watterberg, MD, Principal Investigator — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas Southwestern Medical Center at Dalla; Jon E Tyson, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Eric Eichenwald, MD, Principal Investigator — University of Pennsylvania; Carl T D'Angio, MD, Principal Investigator — University of Rochester; Pablo Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; Bradley Yoder, MD, Principal Investigator — University of Utah
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov)

REFERENCES:
- [Derived] Faix RG, Laptook AR, Shankaran S, Eggleston B, Chowdhury D, Heyne RJ, Das A, Pedroza C, Tyson JE, Wusthoff C, Bonifacio SL, Sanchez PJ, Yoder BA, Laughon MM, Vasil DM, Van Meurs KP, Crawford MM, Higgins RD, Poindexter BB, Colaizy TT, Hamrick SEG, Chalak LF, Ohls RK, Hartley-McAndrew ME, Dysart K, D'Angio CT, Guillet R, Kicklighter SD, Carlo WA, Sokol GM, DeMauro SB, Hibbs AM, Cotten CM, Merhar SL, Bapat RV, Harmon HM, Sewell E, Winter S, Natarajan G, Mosquera R, Hintz SR, Maitre NL, Benninger KL, Peralta-Carcelen M, Hines AC, Duncan AF, Wilson-Costello DE, Trembath A, Malcolm WF, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Whole-Body Hypothermia for Neonatal Encephalopathy in Preterm Infants 33 to 35 Weeks' Gestation: A Randomized Clinical Trial. JAMA Pediatr. 2025 Apr 1;179(4):396-406. doi: 10.1001/jamapediatrics.2024.6613. PMID 39992674
- See also: Neonatal Research Network website — http://neonatal.rti.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole-body Hypothermia | Normothermia
Started | 88 | 80
Completed | 85 | 71
Not Completed | 3 | 9
Not completed — Lost to Follow-up | 3 | 7
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole-body Hypothermia | Normothermia | Total
Number analyzed (Participants) | 88 | 80 | 168
Age, Continuous [Mean (Standard Deviation); unit: Hours] | 4.5 (1.2) | 4.5 (1.3) | 4.5 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 35 | 77
  Male | 46 | 45 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 25
  Not Hispanic or Latino | 71 | 67 | 138
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 31 | 58
  White | 52 | 42 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 88 | 80 | 168
Level of Encephalopathy [Count of Participants; unit: Participants]
  Moderate | 61 | 57 | 118
  Severe | 27 | 23 | 50
Birthweight [Mean (Standard Deviation); unit: grams] | 2463.5 (634.3) | 2371.4 (607.9) | 2419.6 (621.7)
Length [Mean (Standard Deviation); unit: cm] | 46.0 (3.2) | 45.1 (2.8) | 45.6 (3.1)
Gestational Age [Mean (Standard Deviation); unit: Weeks] | 34.0 (0.8) | 34.1 (0.8) | 34 (.8)

OUTCOME MEASURES:

1. Primary Outcome: Death or Moderate or Severe Disability
Description: Severe disability was defined by any of the following: a Bayley III cognitive score < 70 or Gross Motor Function (GMF) Level of 3-5 blindness or profound hearing loss requiring amplification but still unable to following commands/communicate. Moderate disability was defined as a Bayley III cognitive score between 70-84 and either a GMF level of 2 or a seizure disorder or a hearing deficit.
Time Frame: Birth to 18-22 months corrected age
Population: Includes all infants with primary outcome. Does not include 10 lost to follow up, 4 infants without outcome because the Bayley test was not completed, and 2 infants who withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 83 | 69
Participants | 29 | 20
Statistical Analysis 1: Comparison: Whole-body Hypothermia vs Normothermia; Whole-body Hypothermia vs. Normothermia (Normothermia is the comparison group); Test type: Superiority — This trial estimated the probability that the intervention has no effect on the outcome (or conversely, the probability that id does), given the data obtained in the trial and any prior evidence; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.74 to 2.00] — The relative risk estimate was calculated by dividing risk under hypothermia by risk under normothermia; To get estimates of RR from the Bayesian logistic regression model, predicted probabilities of the outcome were generated for all infants assuming the infants were treated with and without hypothermia and with/without severe encephalopathy. Next subject level RR values were estimated for all infants and 2.5, 50, and 97.5 percentiles were calculated

2. Secondary Outcome: Number of Deaths in the NICU and Following Discharge
Description: Number of deaths in the NICU and following discharge among infants with a primary outcome.
Time Frame: Birth to 18-22 months corrected age
Population: Includes all infants with primary outcome. Does not include 10 lost to follow up and 2 infants who withdrew from the study. Also excluded 4 infants without primary outcome because the Bayley test was not completed, so results can be compared with primary outcome which includes death. These 4 infants without primary outcome because the Bayley test was not completed are in the all-cause mortality summary in the Adverse Events module.
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 83 | 69
Participants | 18 | 9

3. Secondary Outcome: Number of Infants With Abnormal MRIs During Post-intervention Period
Description: An MRI was considered abnormal if any abnormal findings were indicated on the CRF form.
Time Frame: Post-intervention to through discharge, death, or transfer (whichever comes first), average of 29 days
Population: Infants who had at least one MRI post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 75 | 67
Participants | 48 | 50

4. Secondary Outcome: Number of Infants With Moderate or Severe Disability
Description: Number of infants with moderate or severe disability among survivors through 18-22 months corrected age.
Time Frame: Birth to 18-22 months corrrected age
Population: infants who were alive at 18-22 months corrected age.
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 65 | 60
Participants | 11 | 11

5. Secondary Outcome: Causes of Death
Description: Causes of any deaths that occurred through 18-22 months corrected age.
Time Frame: Birth to 18-22 months corrrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 18 | 9
Participants
  Asphyxial Brain Injury | 14 | 4
  Multi-organ Failure | 2 | 2
  Cardiomyopathy | 1 | 0
  Complications of HIE | 1 | 0
  BPD/CLD | 0 | 1
  Secondary to severe HIE | 0 | 1
  Pulmonary Hypoplasia | 0 | 1

6. Secondary Outcome: Neurological Injury by Cranial Ultrasound During Intervention
Description: Infants with recorded events of intraventricular hemorrhage grade I, II, III, or IV, posterior fossa hemorrhage with/without shift of midline structures, intraparenchymal hemorrhage.
Time Frame: Within 6 hours of life to 72 hours after start of intervention
Population: Infants who had at least one cranial ultrasound during intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 74 | 67
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs were collected up to 108 hours after baseline. All-cause mortality was collected until 18-22 months corrected age.
Description: SAEs and Other AEs were collected up to 108 hours after baseline. Two randomized infants who withdrew prior to initiation of treatment are excluded from SAE and other AE counting.
Arm/Group | Whole-body Hypothermia | Normothermia
All-Cause Mortality (participants affected / at risk) | 18/88 | 9/80
Serious Adverse Events (participants affected / at risk) | 29/88 | 17/78
Other Adverse Events (participants affected / at risk) | 22/88 | 12/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole-body Hypothermia (N=88) | Normothermia (N=78)
Arrhythmia needing treatment (Cardiac disorders) | 1 (2) | 0 (0)
Intracranial bleeding (Nervous system disorders) | 4 (4) | 4 (4)
Persistent metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (10) | 9 (12)
Major Bleeding (Vascular disorders) | 1 (1) | 4 (4)
Cyanosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PPHN (Congenital, familial and genetic disorders) | 4 (4) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Asphyxial Brain Injury (Nervous system disorders) | 2 (2) | 0 (0)
DIC (General disorders) | 1 (1) | 0 (0)
Death - withdrawal of support (Surgical and medical procedures) | 1 (1) | 0 (0)
Death secondary to severe HIE (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic Cardio-Myopathy (Cardiac disorders) | 1 (1) | 0 (0)
HIE (Nervous system disorders) | 1 (1) | 2 (2)
HIE HYPOXIC ISCHEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
HIE with out come of Death (Nervous system disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Illeal perforation; small bowl resectioned (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neonatal Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neonatal insult (Nervous system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Severe HIE (Nervous system disorders) | 1 (1) | 0 (0)
Severe hypoxic ischemic brain (Nervous system disorders) | 1 (1) | 0 (0)
Spontaneous intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Withdrawal of Support/Death (Surgical and medical procedures) | 1 (1) | 0 (0)
hyperphosphatemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypoxic-ischemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
multiorgan failure and withdrawl of support (Surgical and medical procedures) | 1 (1) | 0 (0)
pleural effusion/pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole-body Hypothermia (N=88) | Normothermia (N=78)
Arrhythmia needing treatment (Cardiac disorders) | 0 (0) | 1 (1)
Persistent metabolic acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Intracranial bleeding (Nervous system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
PPHN (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (15) | 8 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Bilateral mIneralizing vasculopathy (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT01793129/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT01793129/SAP_001.pdf
  • Informed Consent Form (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT01793129/ICF_002.pdf